CLINICAL TRIAL: NCT04770532
Title: A 26-week Trial Comparing the Effect and Safety of Once Weekly Insulin Icodec and Once Daily Insulin Degludec, Both With or Without Non-insulin Anti-diabetic Drugs, in Subjects With Type 2 Diabetes Treated With Basal Insulin
Brief Title: A Research Study to Compare Two Types of Insulin, a New Weekly Insulin, Insulin Icodec and an Available Daily Insulin, Insulin Degludec, in People With Type 2 Diabetes Who Use Daily Insulin
Acronym: ONWARDS 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4478; U1111-1247-4945 (Other: World Health Organization (WHO)); 2020-000454-10 (EudraCT Number)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec; insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin icodec (Experimental): Insulin icodec + non-insulin anti-diabetic drugs. Pre-trial non-insulin anti-diabetic background medication throughout the entire trial except from sulfonylureas and glinides, which must be discontinued at randomisation. The background medication should be maintained at the stable, pre-trial dose and at the same frequency during the entire treatment period.
  Interventions: Drug: Insulin Icodec
- Insulin degludec (Active Comparator): Insulin degludec + non-insulin anti-diabetic drugs. Pre-trial non-insulin anti-diabetic background medication throughout the entire trial except from sulfonylureas and glinides, which must be discontinued at randomisation. The background medication should be maintained at the stable, pre-trial dose and at the same frequency during the entire treatment period.
  Interventions: Drug: Insulin degludec

INTERVENTIONS:
Drug: Insulin degludec — Participants will receive subcutaneous (s.c.) injections of insulin degludec once daily for 26 weeks
  Arms: Insulin degludec
Drug: Insulin Icodec — Participants will receive subcutaneous (s.c.) injections of insulin icodec once weekly for 26 weeks
  Arms: Insulin icodec

SUMMARY:
This study compares insulin icodec (a new insulin taken once a week) to insulin degludec (an insulin taken once daily which is already available on the market) in people with type 2 diabetes.

The study will look at how well insulin icodec taken weekly controls blood sugar compared to insulin degludec taken daily. Participants will either get insulin icodec that participants will have to inject once a week on the same day of the week or insulin degludec that participants will have to inject once a day at the same time every day. Which treatment participants get is decided by chance.

The insulin is injected with a needle in a skin fold in the thigh, upper arm or stomach.

The study will last for about 8 months. Participants will have 17 clinic visits and 13 phone calls with the study doctor. At 8 clinic visits participants will have blood samples taken. At 4 clinic visits participants cannot eat or drink (except for water) for 8 hours before the visit.

Participants will be asked to wear a sensor that measures their blood sugar all the time in 3 periods for a total of 13 weeks (about 3 months) during the study.

Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged above or equal to 18 years at the time of signing informed consent.
* Diagnosed with T2D greater than or equal to 180 days prior to the day of screening.
* HbA1c from 7.0-10.0% (53.0 85.8 mmol/mol) both inclusive at screening confirmed by central laboratory analysis.
* Treated with once daily or twice daily basal insulin (Neutral Protamine Hagedorn insulin, insulin degludec, insulin detemir, insulin glargine 100 units/mL, or insulin glargine 300 units/mL): greater than or equal to 90 days prior to the day of screening with or without any of the following anti-diabetic drugs/regimens with stable doses greater than or equal to 90 days prior to screening:

  * Metformin
  * Sulfonylureas
  * Meglitinides (glinides)
  * DPP-4 inhibitors
  * SGLT2 inhibitors
  * Thiazolidinediones
  * Alpha-glucosidase inhibitors
  * Oral combination products (for the allowed individual oral anti-diabetic drugs)
  * Oral or injectable GLP-1-receptor agonists
* Body mass index (BMI) below or equal to 40.0 kg/m^2.

Exclusion Criteria:

* Any episodes (as declared by the subject or in the medical records) of diabetic ketoacidosis within 90 days prior to the day of screening.
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening.
* Chronic heart failure classified as being in New York Heart Association Class IV at screening.
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or corticosteroids).
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (88):
- United States (38):
  - American Clinical Trials, Buena Park, California
  - Cedars-Sinai Medical Group, Encino, California
  - Valley Research, Fresno, California
  - Diabetes/Lipid Mgmt & Res Ctr, Huntington Beach, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - Clinical Trials Research_Sacramento, Lincoln, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - South Broward Research LLC, Miramar, Florida
  - Renstar Medical Research, Ocala, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endo Res Solutions Inc, Roswell, Georgia
  - Velocity Clin. Res Valparaiso, Valparaiso, Indiana
  - Four Rivers Clinical Research Inc, Paducah, Kentucky
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Ileana J Tandron APMC, Slidell, Louisiana
  - Endo And Metab Cons, Rockville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - MassResearch, LLC, Waltham, Massachusetts
  - Palm Research Center Inc., Las Vegas, Nevada
  - AMC Community Endocrinology, Albany, New York
  - Northport VA Med Ctr Northport, Northport, New York
  - Mountain Diabetes & Endocrine Center, Asheville, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Osvaldo A. Brusco MD PA, Corpus Christi, Texas
  - Thyroid, Endocrinology, and Diabetes, PA, Dallas, Texas
  - Baylr Sctt White Rs Inst, Endo, Dallas, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Diabetes and Thyroid Ctr of FW, Fort Worth, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Capital Clin Res Ctr,LLC, Olympia, Washington
- Bulgaria (6):
  - Medical center Medi City 21 OOD, Kyustendil
  - MHAT Med Line Clinic, Plovdiv
  - OCIPSOMCEMD ENDO MED-CONSULT - Dr. Nikolay Botushanov, Plovdiv
  - ASOMCEM - Individual Practice - Dr. Antoanela Slavcheva, Rousse
  - MMA-MHAT Sofia, Clinic of Endocrinology and Metab. Diseases, Sofia
  - UMHAT Sofiamed EAD, Sofia
- Germany (8):
  - InnoDiab Forschung GmbH, Essen
  - Wendisch/Dahl Hamburg (DZHW), Hamburg
  - Milek, Hohenmölsen, Hohenmölsen
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - Praxis Dr. med. Wenzl-Bauer, Rehlingen-Siersburg
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
  - VvP Kliniken gGmbH Marienhospital Stuttgart - Innere Medizin I, Stuttgart
  - MZM Praxis Drs. Erlinger, Stuttgart
- Japan (9):
  - Hayashi Diabetes Clinic_Internal Medicine and Diabetes Medicine, Chigasaki-shi, Kanagawa, Japan
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - Tokuyama clinic_Diabetic internal medicine, Chiba
  - Futata Tetsuhiro Clinic Meinohama_Internal medicine, Fukuoka-shi, Fukuoka
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Yuri Ono Clinic, Sapporo-shi, Hokkaido
  - Oyama East Clinic_Internal Medicine, Tochigi
  - Juntendo University Hospital_Tokyo, Tokyo
  - Noritake Clinic, Ushiku-shi, Ibaraki
- Poland (3):
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - NZOZ "DiabMed" Poradnia Diabetologiczna, Poznan
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
- Portugal (7):
  - Unidade Local De Saude De Matosinhos E.P.E., Senhora Da Hora, Matosinhos, Matosinhos
  - Unidade Local De Saude De Almada-Seixal E.P.E. - Hospital Garcia de Orta, Almada
  - Unidade Local de Saúde de Coimbra, E.P.E., Coimbra
  - Unidade Local De Saude De Lisboa Ocidental E.P.E. - Hospital Egas Moniz, Lisbon
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - Unidade Local de Saude de Sao Joao E.P.E, Porto
  - Hospital Luz Arrabida, S.A., Vila Nova de Gaia
- South Africa (6):
  - Greenacres Hospital, Port Elizabeth, Eastern Cape
  - Medi-Clinic Bloemfontein, Bloemfontein, Free State
  - Hemant Makan, Johannesburg, Gauteng
  - Chris Hani Baragwanath Hospital, Johannesburg, Gauteng
  - Centre for Diabetes, Johannesburg, Gauteng
  - Dr A Amod, Durban, KwaZulu-Natal
- South Korea (7):
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
- Ukraine (4):
  - "University Clinic" of Dnipro State Medical University - Endocrinology department, Dnipro
  - Department of Medical Service and Rehabilitation of "ARTEM" - day hospital department, Kyiv
  - Komisarenko Institute of Endocrinology and Metabolism of NAMSU - Department of paediatric endocrine pathology, Kyiv
  - Ternopil Central District Hospital - Outpatient department, Ternopil

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Philis-Tsimikas A, Bajaj HS, Begtrup K, Cailleteau R, Gowda A, Lingvay I, Mathieu C, Russell-Jones D, Rosenstock J. Rationale and design of the phase 3a development programme (ONWARDS 1-6 trials) investigating once-weekly insulin icodec in diabetes. Diabetes Obes Metab. 2023 Feb;25(2):331-341. doi: 10.1111/dom.14871. Epub 2022 Oct 14. PMID 36106652
- [Result] Philis-Tsimikas A, Asong M, Franek E, Jia T, Rosenstock J, Stachlewska K, Watada H, Kellerer M. Switching to once-weekly insulin icodec versus once-daily insulin degludec in individuals with basal insulin-treated type 2 diabetes (ONWARDS 2): a phase 3a, randomised, open label, multicentre, treat-to-target trial. Lancet Diabetes Endocrinol. 2023 Jun;11(6):414-425. doi: 10.1016/S2213-8587(23)00093-1. Epub 2023 May 3. PMID 37148899
- [Derived] Philis-Tsimikas A, Krogsdahl Bache J, Fu A, Kellerer M, Salvesen-Sykes K, Bain SC. Insights on Hospitalisations from the Phase 3a ONWARDS 1-6 Trials of Once-Weekly Insulin Icodec. Diabetes Ther. 2025 Aug;16(8):1615-1631. doi: 10.1007/s13300-025-01745-4. Epub 2025 Jun 4. PMID 40465144
- [Derived] Riddell MC, Heller S, Carstensen L, Rocha TMP, Kehlet Watt S, Woo VC. The effect of once-weekly insulin icodec vs once-daily basal insulin on physical activity-attributed hypoglycaemia in type 2 diabetes: a post hoc analysis of ONWARDS 1-5. Diabetologia. 2025 Jul;68(7):1416-1422. doi: 10.1007/s00125-025-06414-6. Epub 2025 Apr 5. PMID 40186685
- [Derived] Polonsky W, Benamar M, Carstensen L, Davies M, Meller Donatsky A, Franek E, Kellerer M, Philis-Tsimikas A, Goldenberg R. Improved treatment satisfaction with once-weekly insulin icodec compared with once-daily basal insulin in individuals with type 2 diabetes: An analysis of patient-reported outcomes and participant interviews from ONWARDS 2 and 5 and a physician survey from ONWARDS 1. Diabetes Res Clin Pract. 2024 Nov;217:111885. doi: 10.1016/j.diabres.2024.111885. Epub 2024 Oct 4. PMID 39368488
- [Derived] Watada H, Asbjornsdottir B, Nishida T, Nishimura R, Yamamoto Y, Yamauchi T, Kadowaki T. Efficacy and safety of once-weekly insulin icodec versus once-daily basal insulin in Japanese individuals with type 2 diabetes: A subgroup analysis of the ONWARDS 1, 2 and 4 trials. Diabetes Obes Metab. 2024 Dec;26(12):5882-5895. doi: 10.1111/dom.15960. Epub 2024 Sep 30. PMID 39344833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 71 sites in 9 countries as follows: United States of America (USA) (26), Ukraine (4), Portugal (6), Poland (3), Republic of Korea (7), Japan (9), Germany (6), Bulgaria (4), South Africa (6).
Pre-assignment Details: After randomisation participants continued their pre-trial non-insulin anti-diabetic background medication throughout the entire trial except from sulfonylureas and glinides, which had to be discontinued at randomisation.
Groups:
- Insulin Icodec: Participants were to receive once weekly subcutaneous (s.c.) injection of Insulin icodec for 26 weeks, using PDS290 prefilled pen-injector at a starting dose of 7 times the pre-trial total daily basal insulin dose + 50% of their 7 times total daily basal insulin dose. The following weekly dose was 7 times the total daily dose of the respective participants ('unit to unit switch' approach: current daily dose x 7). Participants were to perform once daily pre-breakfast self-monitoring plasma glucose (SMPG). The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 millimoles per liter (mmol/L): dose reduced by 3 units (U); 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: dose increased by 3 U.
- Insulin Degludec: Participants were to receive once daily s.c. injection of Insulin degludec for 26 weeks, using PDS290 prefilled pen-injector at a dose in accordance with local label. Participants were to perform once daily SMPG. The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 mmol/L: dose reduced by 20 U; 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: dose increased by 20 U.
Period: Overall Study
Arm/Group | Insulin Icodec | Insulin Degludec
Started | 263 | 263
Exposed | 262 | 263
Full Analysis Set (FAS) | 263 | 263
Safety Analysis Set (SAS) | 262 | 263
Completed | 260 | 258
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Death | 2 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Icodec | Insulin Degludec | Total
Number analyzed (Participants) | 263 | 263 | 526
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.35 (9.79) | 62.60 (8.42) | 62.47 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 123 | 224
  Male | 162 | 140 | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 32
  Not Hispanic or Latino | 247 | 247 | 494
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 86 | 110 | 196
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
  Black or African American | 11 | 12 | 23
  White | 161 | 137 | 298
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline week 0 to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 263 | 263
Percentage of HbA1c | -0.93 (0.05) | -0.71 (0.06)
Statistical Analysis 1: Comparison: Insulin Icodec vs Insulin Degludec; The response and change from baseline in response after 26 weeks were analysed using an analysis of covariance (ANCOVA) model with treatment, region and personal continuous glucose monitoring (CGM) device use as fixed factors, and baseline response as covariate; Test type: Non-Inferiority — Non-inferiority of insulin icodec was considered confirmed if the upper limit of the two-sided 95% confidence interval (CI) for mean treatment difference (insulin icodec minus insulin degludec) was strictly below 0.3%; p < 0.0001, ANCOVA; Treatment difference = -0.22, 95% CI 2-sided [-0.37 to -0.08]

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline week 0 to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all randomised participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 260 | 257
millimoles per liter (mmol/L) | -1.58 (0.12) | -1.62 (0.12)

3. Secondary Outcome: Percentage of Time in Target-range 3.9-10.0 Millimoles Per Liter (mmol/L) (70-180 Milligrams Per Deciliter [mg/dL]) Using Continuous Glucose Monitoring (CGM) System
Description: The percentage of time in target-range 3.9-10.0 mmol/L (70-180 milligrams per deciliter [mg/dL]) using continuous glucose monitoring (CGM) system is presented. Time in target range is defined as 100 times the number of recorded measurements in glycaemic target range 3.9-10.0 mmol/L (70-180 mg/dL), both inclusive, divided by the total number of recorded measurements. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: From week 22 to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage (%) of time
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 238 | 239
Percentage (%) of time | 63.13 (17.40) | 59.50 (18.92)

4. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQs) in Total Treatment Satisfaction
Description: Change in DTSQs in total treatment satisfaction from baseline (week 0) to week 26 is presented. The DTSQ domain score in total treatment satisfaction was calculated by adding the six item scores of items 1, 4-8. Higher scores indicate higher levels of treatment satisfaction for items 1, 4 -8. For items 2 and 3 a higher score indicates a participant perceived experience of hyperglycaemia and hypoglycaemia. Lower scores indicate a perception of blood glucose levels being unacceptably high (item 2) or low (item 3). The score has a minimum of 0 and a maximum of 36. The outcome data was evaluated based on in-trial observation period. In-trial observation period started at randomisation and ended at the date of: Last direct participant-site contact, withdrawal for participants who withdrew their informed consent, last participant-investigator contact as defined by the investigator for participants who were lost to follow-up and death for participants who died before any of the above.
Time Frame: Baseline (Week 0), Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 252 | 244
Score on a scale | 4.22 (0.30) | 2.96 (0.31)

5. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Number of severe hypoglycaemic episodes (level 3) is presented. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. The outcome data was evaluated based on the on-treatment observation period. The on-treatment period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit (V30), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period. The on-treatment period represented the time period in which a participant was considered exposed to trial product.
Time Frame: From baseline (week 0) to week 31
Population: Safety analysis set included all participants randomly assigned to trial treatment and who took at least 1 dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 262 | 263
Episodes | 0 | 1

6. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter)
Description: Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by blood glucose (BG) meter) is presented. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL) confirmed by BG meter. The outcome data was evaluated based on the on-treatment observation period. The on-treatment period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit (V30), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period. The on-treatment period represented the time period in which a participant was considered exposed to trial product.
Time Frame: From baseline (week 0) to week 31
Population: as for outcome 5
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 262 | 263
Episodes | 113 | 41

7. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by blood glucose (BG) meter) or severe hypoglycaemic episodes (level 3) is presented. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of < 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. The outcome data was evaluated based on the in-trial observation period. The on-treatment period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit (V30), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period.
Time Frame: From baseline (week 0) to week 31
Population: as for outcome 5
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 262 | 263
Episodes | 113 | 42

8. Secondary Outcome: Percentage of Time Spent < 3.0 mmol/L (54 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of tiime spent < 3.0 millimoles per liter (mmol/L) (54 mg/dL) using continuous glucose monitoring (CGM) system is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: From week 22 to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage (%) of time
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 238 | 239
Percentage (%) of time | 0.34 (0.88) | 0.22 (0.45)

9. Secondary Outcome: Percentage of Time Spent > 10 mmol/L (180 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time spent > 10 millimoles per liter (mmol/L) (180 milligrams per deciliter [mg/dL]) using continuous glucose monitoring (CGM) system is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: From week 22 to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage (%) of time
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 238 | 239
Percentage (%) of time | 35.52 (17.95) | 39.71 (19.34)

10. Secondary Outcome: Mean Weekly Insulin Dose
Description: Estimated mean weekly insulin dose during the last 2 weeks of treatment (from week 24 to week 26) is presented. The outcome data was evaluated based on the on-treatment observation period. The on-treatment period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: The end of trial visit (V30), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin (corresponding to 5 weeks after the end of the dosing interval for both treatment arms) and the end-date for the in-trial observation period. The on-treatment period represented the time period in which a participant was considered exposed to trial product.
Time Frame: From week 24 to week 26
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units of insulin
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 263 | 263
Units of insulin | 267.96 [252.19 to 284.70] | 244.22 [229.99 to 259.33]

11. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline week 0 to week 26 is presented. The outcome data was evaluated based on the in-trial observation period. In-trial observation period started at randomisation and ended at the date of: The last direct participant-site contact, withdrawal for participants who withdrew their informed consent, the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e., possibly an unscheduled phone visit) and death for participants who died before any of the above.
Time Frame: Baseline (Week 0), Week 26
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | Insulin Icodec | Insulin Degludec
Number analyzed (Participants) | 263 | 263
Kilograms (kg) | 1.40 (0.32) | -0.30 (0.36)

ADVERSE EVENTS:
Time Frame: From baseline (Week 0) to Week 31
Description: All presented adverse events (AEs) are treatment emergent. A treatment-emergent AE (TEAE) was defined as an AE that initiated or worsened on or after the date of first dose of study drug up to the end of the trial period (week 31). Results are based on the safety analysis set which included all randomised participants assigned to trial treatment and who took at least 1 dose of trial product.
Arm/Group | Insulin Icodec | Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 2/262 | 2/263
Serious Adverse Events (participants affected / at risk) | 22/262 | 16/263
Other Adverse Events (participants affected / at risk) | 50/262 | 39/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=262) | Insulin Degludec (N=263)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraspinal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=262) | Insulin Degludec (N=263)
Diabetic retinopathy (Eye disorders) | 10 (11) | 16 (17)
Diarrhoea (Gastrointestinal disorders) | 14 (17) | 9 (9)
Headache (Nervous system disorders) | 14 (20) | 9 (10)
Nasopharyngitis (Infections and infestations) | 22 (28) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04770532/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT04770532/SAP_001.pdf